CLINICAL TRIAL: NCT06804993
Title: Rectocele Repair with or Without Internal Sphincter Botulinum Toxin Injection: a Prospective Randomized Trial
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mostafa shalaby, MD, MSc, PhD, Associate Professor & Consultant Colorectal Surgeon, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MD.21.03.441
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Obstructed Defaecation Syndrome; Anterior Rectocele
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transvaginal repair & botulinum toxin type A toxin injection (Experimental)
  Interventions: Drug: Transvaginal repair & botulinum toxin type A injection
- Transvaginal repair & distilled water injection (Placebo Comparator)
  Interventions: Procedure: Transvaginal repair & distilled water injection

INTERVENTIONS:
Drug: Transvaginal repair & botulinum toxin type A injection — 100 units of lyophilized botulinum toxin type A were diluted in saline to 50 U/mL before the injections. A total of 30 units of type-A botulinum toxin was injected with a 22-G needle evenly divided in 3 sites, 2 on either side of the internal anal sphincter (3 and 9 O'clock) and the third anteriorly (at 12 O'clock)
  Arms: Transvaginal repair & botulinum toxin type A toxin injection
Procedure: Transvaginal repair & distilled water injection — A total of 30 units of distilled water was injected with a 22-G needle evenly divided into 3 sites, 2 on either side of the internal anal sphincter (3 and 9 O'clock) and the third anteriorly (at 12 O'clock)
  Arms: Transvaginal repair & distilled water injection

SUMMARY:
This is a single-centre, prospective randomized controlled trial on female patients with anterior rectocele associated with obstructed defecation syndrome

ELIGIBILITY:
Inclusion Criteria: all required

* female patients
* symptomatic rectocele
* failed conservative treatments for at least 3 months
* anterior rectocele larger than 3 cm in size in defecogram.
* retention of the contrast in the rectocele on defecography
* obstructed defecation manifestations: excessive straining, a sense of incomplete evacuation, the need for digital manipulation during defecation, or dyspareunia

Exclusion Criteria:

* significant urinary manifestations due to anterior vaginal wall prolapse
* recurrent rectocele
* previous anal surgery
* slow-transit constipation
* faecal incontinence (FI)
* abnormal thyroid functions
* patients under systemic steroid treatment
* patients with connective tissue disease
* ASA classification >3

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2021-07-31 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No